CLINICAL TRIAL: NCT01854905
Title: An Observational Study of Dry Eye Prior to Laser-Assisted in Situ Keratomileusis (LASIK) Therapy
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: MAF-AGN-OPH-DE-015
Record Dates: First submitted 2013-05-14; First posted 2013-05-16 (Estimated); Results first posted 2014-03-14 (Estimated); Last update posted 2014-03-14 (Estimated); Status verified 2014-01

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients Attending Consultation for LASIK: Patients attending consultation for LASIK on Day 1. No intervention or treatment is administered during the study.
  Interventions: Other: No Treatment

INTERVENTIONS:
Other: No Treatment — Patients attending consultation for LASIK on Day 1. No intervention or treatment is administered during the study.

SUMMARY:
This is an observational, study of dry eye in patients at the consultation visit prior to LASIK surgery. There is no treatment administered or intervention during the study.

ELIGIBILITY:
Inclusion Criteria:

* Attending an ophthalmology consultation for LASIK

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients consulting with ophthalmologist for possible LASIK
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2013-05; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Moscow, Russia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients Attending Consultation for LASIK
Started | 400
Completed | 400
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients Attending Consultation for LASIK
Number analyzed (Participants) | 400
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.7 (9.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 263
  Male | 137

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients in Each Category of the Dry Eye Workshop Severity (DEWS) Scale
Description: The severity of each patient's dry eye was classified by the physician according to the DEWS scale. Categories are: mild and/or episodic, occurs under environmental stress; moderate episodic or chronic, stress or no stress; and severe frequent or constant without stress
Time Frame: Day 1
Population: All enrolled patients
Measure: Number; unit: Percentage of Patients
Arm/Group | Patients Attending Consultation for LASIK
Number analyzed (Participants) | 400
Percentage of Patients
  Mild and/or episodic, occurs under stress | 65.0 (25.97)
  Moderate episodic or chronic, stress or no stress | 29.0
  Severe frequent or constant without stress | 4.2
  Data unavailable | 1.8

ADVERSE EVENTS:
Description: Adverse events (AEs) and serious adverse events (SAEs) were not collected in this single day study, as no treatment was administered.
Arm/Group | Patients Attending Consultation for LASIK
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.